

# The RELIEF Trial

REstrictive versus LIbEral Fluid Therapy in Major Abdominal Surgery

# www.relief.org.au

On behalf of the Australian and New Zealand College of Anaesthetists Clinical Trials Network (ANZCA CTN), and the Australian and New Zealand Intensive Care Society Clinical Trials Group (ANZICS CTG)

ClinicalTrials.gov Identifier: NCT01424150

Protocol Version 2: 3<sup>rd</sup> August 2016

Study title: Restrictive versus liberal fluid therapy in major abdominal surgery

Protocol Number: Anaesthesia Research 046

Sponsor: Alfred Health, Melbourne

Funding source: The Australian National Health and Medical Research Council (APP1043755)

# **AGREEMENT**

| This document is confidential. The Investigators declare that amendments. The Investigators will conduct the study according accordance with ICH GCP notes for Guidance on Good Clini NH&MRC National Statement on Ethical Conduct in Research | ding to the procedures specified in the study protocol, and cal Practice (CPMP/ICH/135/95) and the Australian |
|---|---|
| Investigator | Date |

# RELIEF: REstrictive versus LIbEral Fluid Therapy in Major Abdominal Surgery

# **Principal Investigator**

Paul Myles, MB.BS, MPH, MD, FCAI, FANZCA, FRCA, FAHMS

Director, Department of Anaesthesia and Perioperative Medicine, Alfred Hospital and Monash University

## **Intensive Care**

Rinaldo Bellomo, MB.BS, MD, FRACP, FCICM, PGDipEcho

Co-Director of the ANZIC-RC and the Director of Intensive Care Research at Austin Health

#### **Anaesthesia**

Tomas Corcoran, MB, BCh, BAO, MRCPI, FCAI, MD, FCICM

Department of Anaesthesia and Pain Medicine, Royal Perth Hospital; School of Medicine and Pharmacology, University of Western Australia

Philip Peyton, MD, PhD, MB.BS, FANZCA, PGDipEcho

Staff Anaesthetist, Department of Anaesthesia, Austin Health

David Story, MBBS, MD, BMedSci, FANZCA

Chair of Anaesthesia; and Head, Centre for Anaesthesia, Perioperative and Pain Medicine; The University of Melbourne

Kate Leslie, MB.BS, MD, M Epi, FANZCA

Staff Anaesthetist, Department of Anaesthesia and Pain Management, Royal Melbourne Hospital; University of Melbourne; Monash University

#### Surgery

Chris Christophi, MB.BS, FRACS

Director of Surgery, Austin Hospital and University of Melbourne

Jonathan Serpell, MB.BS, MD, Med, FRACS, FACS

Director, Department of General Surgery, Alfred Hospital and Monash University

# Statistician

Andrew Forbes MSc, PhD

Head, Biostatistics Unit, Department of Epidemiology & Preventive Medicine, Monash University

Research Manager: Sophie Wallace

# **Data and Safety Monitoring Committee**

Monty Mythen (Chair, *intensivist*, Smiths Medical Professor of Anaesthesia & Critical Care, University College London (UK); Russell Gruen (*surgeon*), Guy Ludbrook (*anaesthetist*), John McNeil (*epidemiologist*), Katherine Lee (*statistician*).

Endpoint Adjudication Committee: David McIlroy, Mark Shulman, Jamie Cooper

Governance and Data Quality Manager: Sophie Wallace

# **ABBREVIATIONS**

ACE - angiotensin converting enzyme

ANZCA TG - Australian and New Zealand College of Anaesthetists Trials Group

ANZICS CTG – Australian and New Zealand Intensive Care Society Clinical Trials Group

APTT – activated partial thromboplastin time

ARB - angiotensin-II receptor blocker

ASA – American Association of Anesthesiologists

ATACAS – Aspirin and Tranexamic Acid for Coronary Artery Surgery trial

BMI - Body Mass Index

BP - Blood Pressure

CXR - Chest X-Ray

CRF - Case Report Form

CT - computed tomography scan

CVP - Central Venous Pressure

CD - Compact Disc

CDC - Centers for Disease Control and Prevention

CRP - C-reactive protein

DO2 – Tissue oxygen delivery

DSMC - Data Safety and Monitoring Committee

EAC - Endpoint Adjudication Committee

ECG - Electrocardiography

ENIGMA - Evaluation of Nitrous Oxide in the Gas mixture for Anaesthesia

ENIGMA-II - Nitrous oxide anaesthesia and cardiac morbidity after major surgery

ERAS - Enhanced Recovery After Surgery

FiO2 - Fraction of Inspired Oxygen

FTc - Flow Time Corrected

GA - General Anaesthesia

GCP - Good Clinical Practice

GFR - Glomerular filtration Rate

HR - Heart Rate

HDU – High Dependency Unit

INR - International Normalized Ratio

ICP - Intracranial Pressure

ICU - Intensive Care Unit

IV - Intravenous

IVRS – Interacive Voice Response System

L - Litres

PRN - as the occasion arises; as needed.

RIFLE - Risk, Injury, Failure, Loss, and End-stage kidney classification

NHMRC - Australian National Health and Medical Research Council

NHSN - National Healthcare Safety Network

mmol/L - Millimole per Litre

mmHg - millimetres of mercury

OR – Operating Room

PA - Pulmonary Artery

PaO2 – Arterial partial pressure of oxygen

PI&CF - Patient Information and Consent form

PPV - Positive Pressure Ventilation

QoR-40 - 40-item Quality of Recovery score

SAFE - Saline versus Albumin Fluid Evaluation study

sBP - Systolic Blood Pressure

SVV - Stroke Volume Variation

TGA – Australian Therapeutic Goods Administration

TOE - transoesophageal echocardiography, or TEE

WCC - White Cell Count

WHODAS - World Health Organization Disability Assessment Schedule

#### **TRIAL SUMMARY**

**Design**: This will be a large, randomized, parallel-group, controlled trial. After stratification by centre *and* planned ICU/HDU admission (or not), patients will be randomly assigned from a computer-generated list (1:1) to either a Restrictive or Liberal fluid Group.

**Group 1** = Restrictive fluid regimen (intraoperative and  $1^{st}$  24 h ≈2.5 L) **Group 2** = Liberal fluid regimen (intraoperative and  $1^{st}$  24 h ≈5.5 L)

Sample Size: 3000 patients

Study Duration: 3 years

#### **Primary Endpoint**

Disability-free survival up to 1 year: survival and freedom from disability after surgery, the latter being a persistent (>6 months) reduction in functional status as defined by a 4-point or greater reduction in the 12-item version of WHODAS. Disability will be assessed by the participant, but if unable then we will use the proxy's report. The date of onset of new disability will be recorded.

Interim analysis (& DSMC review): at n≈ 1500 patients

#### 1. AIM OF THE TRIAL

To investigate the effectiveness of fluid restriction (vs. liberal), and the possible effect-modification of goal-directed therapy (eg. oesophageal Doppler, Flotrac®). The first will be randomly assigned; the latter will be measured covariates according to local practices and beliefs.

The optimal fluid regimen and haemodynamic (or other) targets for patients undergoing major surgery are based on rationales that are not supported by strong evidence. Practices vary substantially; guidelines are vague, small trials and meta-analyses are contradictory. The strongest and most consistent evidence, and biological plausability regarding tissue oedema, supports a restrictive fluid strategy. There is less (and more contradictory) evidence supporting goal-directed therapy using a flow-directed device and/or dopexamine, and use and choice of colloids. A large, definitive clinical trial evaluating perioperative fluid replacement in major surgery is required.

# 1.1 Study Hypotheses

A restrictive fluid regimen for adults undergoing major abdominal surgery leads to reduced complications and improved disability-free survival when compared with a liberal fluid regimen.

Secondary hypotheses: The effects of fluid restriction are similar whether or not goal-directed therapy is used (assessed as a statistical test of interaction). A restrictive fluid regimen will reduce a composite of 30-day septic complications and mortality.

#### 2. BACKGROUND

Anaesthetists typically manage perioperative hypotension in the first instance with an intravenous (IV) fluid bolus of a balanced salt crystalloid solution, or sometimes with one of several colloids. If persistent or more profound hypotension occurs, particularly in the intraoperative period when anaesthetic drug-induced vasodilation is common, an IV vasoconstrictor (typically metaraminol bolus prn) is used. Similar approaches are used in the intensive care unit (ICU) and surgical wards. We simply don't know whether using a 'liberal' fluid strategy based primarily on supplemental IV fluids, or a 'restrictive' strategy based on altered haemodynamic goals and/or vasopressor drug therapy, is best for most patients undergoing major surgery. The evidence base for fluid management in the postoperative setting is poor and is insufficient to guide our practice (1-4). Anaesthetists, intensivists and surgeons differ in their approaches to perioperative fluid therapy (5, 6).

Around 250 million people undergo major surgery each year around the world (7), with about 2 million being in Australia (1 in 10 Australians), and a growing proportion (now 40%) being elderly. By 2056 in Australia, more than 8.5 million anaesthetics (>50%) will be administered to patients over the age of 65 (8). These patients and many others have co-existent medical diseases that add risk to the procedure. The personal, social and economic consequences of postoperative complications, additional hospital stay, and long-term disability, are great.

Both colloids and crystalloids are used for fluid resuscitation and maintenance, but it is the amount of fluids administered and the goals of resuscitation that need re-evaluation. Since the 1950s, when it was first claimed that after surgery fluids are redistributed to a theoretical 'third space' (9), perioperative IV fluid replacement has included replacement of such third-space losses with crystalloid. In fact there are many reasons why clinicians administer generous amounts of IV fluids during and after surgery. Concerns about reversing preoperative dehydration, support ingthe circulation after general and regional anaesthesia, avoiding gut hypoperfusion and promoting tissue oxygen delivery, avoiding blood transfusion, and maintaining urine output are common (10-12). Optimizing tissue perfusion typically requires more fluid than indicated by normal clinical criteria or with invasive monitoring (10). Occult hypovolaemia and intraoperative gut hypoperfusion occurs in around 60% of major surgery patients, both of which are linked to increases in morbidity and mortality (11). Further support for this comes from some studies showing that a liberal fluid strategy in patients undergoing minor surgery, mostly in the ambulatory setting, improves early recovery measures such as dizziness, nausea and thirst, and may improve pulmonary function, exercise capacity, and shorten hospital stay (13). Similarly in the ICU setting, with some small trials suggest that fluid supplementation and optimized haemodynamics reduce organ dysfunction, postoperative morbidity and death (14, 15).

If fluid administration is restricted it is likely that hypotension will be treated with vasopressor therapy. Vasopressors may impair organ perfusion, threaten local tissues at the site of IV administration, cause arrhythmias, or be mistakenly used when hypovolaemia is the underlying cause.

But excess fluid administration causes oedema, with increased pulmonary morbidity (16), impaired coagulation (17), bacterial translocation and sepsis (18), and poor wound healing. In contrast to the above, other small trials of patients undergoing abdominal surgery have found that fluid restriction lead to reduced morbidity and hospital stay (12, 13). This conflicting evidence explains why there are diverse and varied practices around the world. Several expert guideline/consensus statements have been published, with most supporting restrictive fluid administration (2, 19). But all come to similar conclusions: High-grade evidence regarding the optimal fluid regimen is currently lacking (19).

# 2.1 Liberal or Restrictive IV Fluid Resuscitation

Traditional perioperative IV fluid regimens in abdominal surgery can lead to patients receiving 3 to 7 L of fluid on the day of surgery and more than 3 L/day for the following 3 to 4 days, leading to a 3- to 6-kg weight gain (20, 21). Several small trials have compared restrictive and liberal fluid regimens (3, 22).

Lobo et al (20) did a tightly-controlled randomized trial in 20 adult patients having colonic surgery. The liberal group, representing 'standard' care, received IV fluids in accordance with their present hospital practice (≥3 L/day) and the restrictive group received ≤2 L water and sodium 77 mmol per day. All patients had no comorbidity other than colonic cancer. The restrictive group had shorter median gastric emptying times, less complications (0 vs. 7, P=0.01) and shorter hospital stay (6 vs. 9 days, P=0.001). Brandstrup et al (23) did a randomized trial comparing similar fluid regimens in 172 colorectal surgical patients. The restrictive group had fewer postoperative complications (33% vs. 51%, P=0.013) and less deaths (0 vs. 4, P=0.12). Nisenavich et al (24) compared liberal and restrictive fluid regimens in 152 patients undergoing elective abdominal surgery. The restrictive group had faster return of bowel function, less complications (P=0.046), and shorter hospital stay (P=0.01). Similar benefits were found in recent trials in colorectal and abdominal aortic surgery (25, 26).

However, Kabon et al (25) compared similar fluid regimens in 253 colorectal surgical patients and found no difference in the rates of wound infection, restrictive group 14% vs. liberal group 11% (P=0.46). Holte et al (27) compared two fluid regimens with physiological recovery as the primary outcome measure in 32 patients undergoing fast-track colonic surgery. The rate of complications tended to be higher in the restrictive group (6 vs. 1, P = 0.08). A meta-analysis of the fluid trials up to 2007 (3) found restrictive regimens reduced overall complications, OR 0.41 (95% CI: 0.22-0.77), P=0.005; but the authors noted the heterogeneity of fluid regimens and definitions of outcomes. Another two recent small trials found either no benefit (26) or harm (28).

We have done an updated meta-analysis of relevant trials (12 trials, 1160 patients) to evaluate the overall effect of fluid restriction on mortality (see Fig 1) and some morbidities (22). We could not pool overall complications because of their variability and inconsistency of counting. About half the trials did not measure or report mortality, so this outcome is underpowered. We found some possible benefits of fluid restriction:

- Pneumonia: RR 0.43 (95% CI: 0.20-0.94); P=0.03
- Pulmonary oedema: RR 0.22 (95% CI: 0.06-0.78); P=0.02
- Hospital stay: restrictive groups 2 days less (95% CI: 0.5-3.4); P=0.009
- Hospital mortality: RR 0.59 (95% CI:0.2-2.0); P=0.40

Figure 1. Mortality



Our results show fluid restriction seems very promising and could lead to marked improvements in patient outcomes, but a large definitive trial is needed to generate the reliable evidence needed to change practice around the world.

An earlier meta-analysis that included less relevant trials (4) found that the range of 'liberal' IV fluid replacement varied from 2,750 to 5,388 ml compared with 998 to 2,740 ml in the 'restrictive' regimen. Like others (3) they noted that the fluid regimens and outcomes were inconsistently defined and only two studies reported perioperative care principles and discharge criteria. These and others have argued for a carefully designed trial that incorporates such details.

# 2.2 Crystalloid or Colloid Fluid Resuscitation?

Colloid proponents have argued that colloids lessen the risk of oedema because of the higher oncotic pressure, and textbooks typically recommend a 3-5 fold ratio of crystalloid to colloid volumes for acute fluid resuscitation. But the oncotic pressure effect may be lost if colloids leak and remain in the interstitial spaces. This perhaps explains why recent large trials have found that CVP and pulmonary function are comparable with both crystalloids and colloids (29-31) . The SAFE study found that the volume of crystalloid needed for resuscitation at 24 h was only 1.3-fold larger than that of 4% albumin (32). There is concern regarding the safety of colloids (29-31, 33) .

The weight of evidence downplays the superiority of any particular IV fluid (crystalloid or colloid (32), type of colloid (3), or type of crystalloid. The main unresolved question is how much fluid to use, and whether haemodynamic- or flow-directed goals provide further benefit. However, in view of emerging evidence suggesting adverse effects of starch-based colloid solutions (30, 34), we recommend they NOT be used in this study.

# 2.3 Goal-directed Therapy: fluids and/or inotropes

CVP is an unreliable measure of intravascular status (35), but remains the most common monitor used to guide fluid resuscitation and vasopressor support. Relatively noninvasive monitors such as oesophageal Doppler and pulse contour analysis are becoming popular for intraoperative and ICU use (36), and there have been several positive trials (37-40), meta-analysis (22, 41), and guidelines (42) supporting their use. The strongest evidence is for oesphageal Doppler (42) but the device is infrequently used in Australian practice at present. Goal-directed strategies focus on

fluid responsiveness and typically require additional IV fluid supplementation, usually giving an extra 800 ml per case, and more postoperatively(22). These findings are hard to resolve when considering the apparent success of fluid restriction regimens described above.

One influential trial of 'optimized' care in the UK (15) in which 138 high-risk patients undergoing major abdominal surgery were randomly assigned to one of 3 groups: control, or 'pre-optimized' with either dopexamine or adrenaline. The control group remained on the general surgical ward with no preoperative fluid protocol. The intervention groups were admitted to the ICU for a minimum of 4 h before surgery, and had full haemodynamic monitoring including PA catheter. The two intervention groups were initially fluid optimized with colloid until pulmonary occlusion pressure 12 mm Hg was reached; red cell transfusion was used for haemoglobin <110 g/L. Patients then received inotrope therapy titrated to reach a target DO2 of 600 ml/min/m2 for up to 12±24 h after surgery. Hospital mortality in the protocol groups was 3%, compared with 17% in the control (P=0.007), and morbidity and hospital stay were significantly reduced in the dopexamine group. Interpretation of this study is difficult. It could be said that closer (and more expert) care in the ICU, compared with junior doctor-based ward care, was a key factor. Whether the target DO2 itself, inotrope therapy, additional fluids, or the combination of these factors is important is unclear. Two subsequent meta-analyses of dopexamine in major surgery had conflicting findings (43, 44), and a recent trial using FloTrac-guided fluid supplementation found (45) no effect on complication rate (45).

The most recent meta-analysis (46) of 29 trials involved 4805 patients found pre-emptive perioperative haemodynamic intervention significantly reduced mortality, OR 0.48 [95% CI:0.33–0.78]; P<0.0002; and surgical complications, OR 0.43 [0.34–0.53]; P< 0.0001. That is, supplemental fluids seem to improve outcome. Sub-group analyses showed similar effects with each type of intervention, including use of supplemental IV fluids alone:

| | No. of patients with complications | | | |
|---|---|---|---|---|
| Subgroup | No. of studies | No. of patients | in control group | Odds ratio (95% CI) |
| Monitor | | | | |
| ODM | 9 | 987 | 163/469 (35%) | 0.41 (0.30-0.57)* |
| PAFC | 10 | 1085 | 108/537 (20%) | 0.54 (0.33-0.88)* |
| Other | 4 | 320 | 76/158 (48%) | 0.32 (0.19-0.54)* |
| Therapy | | | | |
| Fluids | 9 | 742 | 126/372 (34%) | 0.38 (0.26-0.55)* |
| Fluids and inotropes | 14 | 1650 | 221/792 (28%) | 0.47 (0.35-0.64)* |
| Goals | | | | |
| CI/Do <sub>2</sub> | 12 | 982 | 169/461 (37%) | 0.52 (0.37-0.74)* |
| FTc/SV | 8 | 849 | 135/423 (32%) | 0.41 (0.28-0.58)* |
| Other <sup>b</sup> | 3 | 561 | 43/280 (15%) | 0.26 (0.13-0.52)* |
| Resuscitation target | | | | |
| Supranormal | 6 | 469 | 133/227 (59%) | 0.42 (0.29-0.63)* |
| Normal | 17 | 1923 | 214/937 (23%) | 0.43 (0.31-0.60)* |

A later trial in 179 patients found no outcome benefit of goal-directed therapy, and possibly longer hospital stay (47).

One of the reasons for the varied results is that the focus should not be on the amount of IV fluid, but the timing and individualisation of such therapy. There may be an optimal amount, probably better targeted using a goal-directed approach (48).

# 2.4 "Fast-track" or "enhanced recovery from surgery" (ERAS) programs

There is a growing interest in facilitating recovery and earlier hospital discharge after colorectal and other abdominal surgery (44-46). ERAS programs typically include avoidance of bowel preparation, nasogastric and drain tubes; non-opioid analgesia; and promoting early postoperative mobilization and oral nutrition. A randomized trial comparing an ERAS program with traditional care in 156 patients undergoing colorectal surgery was stopped early because of apparent benefit (46), with less complications (21% vs. 50%, P=0.001) and a shorter hospital stay (5 vs. 9 days, P<0.001). A regression analysis revealed excess IV fluids (OR 4.2 [95% CI 1.7–10]; P=0.002) as an independent predictor of postoperative complications. A recent meta-analysis of ERAS studies has similarly found a significant reduction in complications and hospital stay (49). Most of the above fluid trials did not employ ERAS principles (4), and so we plan to include these in our study.

# 2.5 Measuring Outcome after Major Abdominal Surgery?

Most of the above-quoted studies pooled a variety of postoperative adverse outcomes into a single composite outcome ("complications"), for which there was often an imbalance in severity and duration, and with questionable long-term relevance to patients. Composite outcomes can be valid and important but only if properly constructed (50). Of course a hard endpoint after surgery is survival, but none of the above studies was sufficiently powered to detect a clinically important difference. Mortality is low after most types of surgery (49, 51) and so is an unattractive primary endpoint on which to base a sample size calculation.

It is unclear which of many adverse postoperative outcomes dominates any other. There is a strong argument to use patient-centred outcome measures. Quality of life is often used, but these instruments were not designed to be responsive after major surgery. Our 40-item quality of recovery score (QoR-40) has undergone psychometric evaluation, including utility and responsiveness testing (51, 52), and has been externally validated and used in many perioperative studies (53-55). But the QoR-40 is designed to measure outcome up to 30 days after surgery. Survival, and avoiding long-term disability, are likely to be the most important and highly valued outcomes for patients undergoing major surgery (56, 57). We thus plan to measure disability-free survival up to 1 year after surgery in this study.

Interim Long-term Outcome Data for ENIGMA-II and ATACAS trials: Our experience to date with 1-year follow-up for death/disability (using Katz ADLs) in our two current large international trials across >30 sites (58, 59) has had excellent follow-up, with <1% missing data (24 of 2,570 patients). For noncardiac surgery (n=1800) there have been 242 deaths and 286 with new disability (a combined rate of 31%). This event rate, from a lower risk study population, exceeds our assumptions used in our sample size calculation. Clearly, disability should not be ignored in perioperative outcome trials, and its inclusion can enhance study power.

#### 2.6 Feasibility: Pilot Study

To ascertain current practices and support for this trial, we surveyed all members of both ANZCA and ANZICS Trials Groups (n=238) and found that >90% were comfortable with the proposed Group fluid regimens and were interested in participating in the trial (60).

We undertook a feasibility pilot study of the proposed trial at 3 centres. After ethics approval and patient consent, and surgeon, anaesthetist and intensivist support, we have demonstrated that we can successfully implement the fluid regimens both intraoperatively and postoperatively:

| variable | Restrictive<br>(n=41) | Liberal<br>(n=41) | P value |
|---|---|---|---|
| Age, y | 65 ± 12 | 67 ± 12 | - |
| IV fluid (crystalloid + colloid) | | | |
| Intraoperative | 1746 ± 748 | 2730 ± 1309 | <0.0005 |
| Total at 24 h postoperative | 3167 ± 1625 | 5133 ± 2138 | <0.0005 |
| Postoperative | | | |
| Haemoglobin, g/L | 110 ± 18 | 101 ± 17 | 0.014 |
| Albumin, g/L | 31 ± 6.7 | 27 ± 7.0 | 0.030 |
| CRP, mg/L | 108 ± 80 | 128 ± 75 | 0.33 |
| Quality of recovery score | 159 ± 20 | 154 ± 26 | 0.34 |
| Median ICU stay, h | 0 (0-15) | 0 (0-19) | 0.86 |
| Median Hospital stay, days | 8.1 (5.6-14) | 8.4 (6.9-16) | 0.30 |

To date there is no evidence of any adverse haemodynamic or renal effects with restrictive therapy (61).

In addition, we are currently undertaking a cohort study of 400 patients undergoing a range of elective surgeries to accurately measure and define rates of comorbidity, wellbeing and disability at 1, 3, 6, and 12 months after surgery. This will validate our follow-up and disability measurement techniques.

#### 3. STUDY DESIGN

#### 3.1 Experimental design

Large, multicentre, randomized, single blind, pragmatic trial, with patients randomly assigned to either Restrictive or Liberal fluid, stratified by site and planned HDU/ICU admission.

This is an effectiveness trial (62, 63) – some elements of the trial are deliberately left to the anaesthetist's discretion in order to reflect usual practice and maximise generalisability.

#### 3.2 Subject Selection

## 3.2.1 Definition of Disease State

We are targeting patients undergoing planned major abdominal or pelvic surgery that includes a skin incision and operative duration expected to exceed two hours.

#### 3.2.2 Source and Number

We will use similar procedures to those used by us successfully in previous multicentre studies. Simple eligibility criteria, and research nurse-screening and enrolment, ensure that recruitment is maximized.

3000 patients in total will be required for this study (1500 in each group).

#### 3.2.3 Entrance Criteria

## Inclusion criteria:

- 1. Adults (≥18 years) undergoing elective major surgery and providing informed consent
- 2. All types of open or lap-assisted abdominal or pelvic surgery with an expected duration of at least 2 hours, and an expected hospital stay of at least 3 days (for example, oesophagectomy, gastrectomy, pancreatectomy, colectomy, aortic or aorto-femoral vascular surgery, nephrectomy, cystectomy, open prostatectomy, radical hysterectomy, and abdominal incisional hernia repair)
- 3. At increased risk of postoperative complications, defined as at least one of the following criteria:
  - a) age ≥70 years
  - b) known or documented history of coronary artery disease
  - c) known or documented history of heart failure
  - d) diabetes currently treated with an oral hypoglycaemic agent and/or insulin
  - e) preoperative serum creatinine >200 μmol/L (>2.8 mg/dl)
  - f) morbid obesity (BMI  $\geq$ 35 kg/m<sup>2</sup>)
  - g) preoperative serum albumin <30 g/L
  - h) anaerobic threshold (if done) <12 mL/kg/min
  - i) or two or more of the following risk factors:
    - ASA 3 or 4
    - chronic respiratory disease
    - obesity (BMI 30-35 kg/m²)
    - aortic or peripheral vascular disease
    - preoperative haemoglobin <100 g/L</li>
    - preoperative serum creatinine 150-199 μmol/L (>1.7 mg/dl)
    - anaerobic threshold (if done) 12-14 mL/kg/min

# Exclusion criteria:

- 1. Urgent or time-critical surgery
- 2. ASA physical status 5 such patients are not expected to survive with or without surgery, and their underlying illness is expected to have an overwhelming effect on outcome (irrespective of fluid therapy)
- 3. Chronic renal failure requiring dialysis
- 4. Pulmonary or cardiac surgery different pathophysiology, and thoracic surgery typically have strict fluid restrictions
- 5. Liver resection most units have strict fluid/CVP limits in place and won't allow randomisation
- **6.** Minor or intermediate surgery, such as laparoscopic cholecystectomy, transurethral resection of the prostate, inguinal hernia repair, splenectomy, closure of colostomy each of these are typically "minor" surgery with minimal IV fluid requirements, generally low rates of complications and mostly very good survival.

#### 3.3 Study Procedures

# 3.3.1 General Description

**Study Flow Chart** 

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | Visit 5 | Visit 6 | Visit 7 | Visit 8 | Visit 9 |
|---|---|---|---|---|---|---|---|---|---|
| | Preadmiss<br>ion Clinic/<br>preoperati<br>ve visit | Day of<br>Surgery | Post op<br>day 1 | Post op day<br>3 | Day of discharge | 30 day<br>follow up<br>phone<br>call | 3 month<br>phone<br>follow-up | 6 month<br>phone<br>follow-up | 12 month<br>phone<br>follow-up |
| Entry Criteria | х | | | | | | | | |
| Informed<br>Consent | x or | r x | | | | | | | |
| Demographics,<br>Medical History | x or | r x | | | | | | | |
| ECG | x or | r x | x | if chest pain or elevated troponin | | roponin | | | |
| Randomisation | | х | | | | | | | |
| Blood tests<br>Electrolytes | x or | r x | х | х | | | | | |
| Liver function tests | If clinically | indicated | If clinically | , indicated | | | | | |
| HbA1C | Recommended in ALL diabetics | | | | | | | | |
| CRP | | | | Х | | | | | |
| Blood tests<br>Troponin<br>Lactate | | If clinically indicated | | | | | | | |
| IV fluids | | х | х | х | | | | | |
| Web-based<br>data entry | | х | | | х | х | х | х | х |
| Wound inspection | | | If change of dressing | х | x | Medical<br>record<br>review | | | |
| QoR-15 | | | х | х | | х | | | |
| WHODAS | Х | | | | | х | х | х | х |
| Adverse Events | | x | x | х | | x | | | |
| Outcomes | | | | | | х | | | |
| Blood products | | х | х | x | х | | | | |

All procedures are based on successful strategies used in each of our previous large multicentre trials. Ethics Committee approval and informed consent will be obtained at all study centres. After enrolment, on the day of surgery, patients will be randomly assigned (1:1) to groups via either (both established) 24-hr freecall telephone or web-based service using a computer-generated code. All other perioperative clinical care will be according to standard practice. All relevant factors will be recorded on a trial case report form (CRF).

# 3.3.2 Perioperative Management

## **Preoperative period**

ERAS perioperative care principles will be emphasized. All patients will receive prophylactic antibiotics according to established guidelines. Medications will be continued perioperatively unless or at the clinicians discretion, but we will recommend withholding ACE-inhibitors and ARBs on the day of surgery. We will record preoperative use of bowel preparation, fasting times, ERAS data, medications, and biochemistry and haematology results on the CRF.

## Intraoperative period

Choice of anaesthetic agents and perioperative analgesia will be left to the discretion of the anaesthetist; such data will be recorded. We will emphasize the need to avoid hypothermia (<36 °C). Epidural use will be recorded as this may

increase the risk of hypotension and need for IV fluids (64, 65), but such effects are likely to be small (66). We will record usage of all "advanced" monitoring devices (CVP, pulse contour analysis, TOE, oesophageal Doppler).

The acceptable limits of low BP, and a definition of 'hypotension', vary widely (67), though such a definition will be modified by older age, pre-existing hypertension, and cerebrovascular disease. We will use a general guideline of systolic BP <90 mmHg for more than 5 mins, but also ask the attending anaesthetist to modify their acceptable lower limit of sBP at the commencement of surgery, and, according to randomly-assigned group, treat hypotension with additional IV fluid or vasopressor therapy (see below). For example, in younger patients or those with pre-existing low BP it may be acceptable to tolerate a sBP of 85-95 mmHg, but in older patients, particularly those with pre-existing hypertension, a higher lower limit may be required. Such modification to the acceptable lower sBP will be recorded. For patients managed in a high dependency or ICU environment after surgery, hypotension will be similarly treated for the first 24 h after surgery.

## Postoperative period

Patients will be followed daily and outcomes will be recorded until discharge. We will recommend that antihypertensive medications should be withheld until sBP is consistently at or above preoperative levels. Serum electrolytes, haemoglobin/haematocrit, and a 12-lead ECG will be ordered preoperatively and on day 1 after surgery. CRP will be measured on postoperative Day 3 and whenever sepsis is suspected (68, 69). Additional laboratory tests will be ordered if clinically indicated. On day 3 all patients will complete the 15-item quality of recovery score (QoR-15). On day 30 all patients will be contacted by phone to ascertain if they have experienced any outcomes, and if detected, further testing will be arranged. Documentation for such events will be sought in the hospital medical record and doctor's records. The QoR-15 will be repeated on day 30 along with WHODAS, and the WHODAS will be repeated at 3-, 6- and 12-month follow-up to ascertain survival status and new-onset disability.

#### 3.3.3 Clinical Observations

#### 3.3.3.1 Primary Endpoint

Disability-free survival up to 1 year: survival and freedom from disability. The latter is defined as a persistent (≥6 months) reduction in health status as measured by a 12-item version of WHODAS (70) score of at least 24 points, reflecting a disability level of at least 25% and being the threshold point between "disabled" and "not disabled" as per WHO guidelines (71). Disability will be assessed by the participant, but if unable then we will use the proxy's report. The date of onset of new disability will be recorded. Further details are provided in the Procedures Manual and the Statistical Analysis Plan.

#### 3.3.3.2 Secondary Endpoints

Secondary endpoints include an *a priori* composite of 30-day mortality or major septic complications (sepsis, surgical site infection, anastomotic leak, and pneumonia), plus each individually, serum lactate (at 6 and 24 h), CRP (Day 3), blood transfusion, acute kidney injury, ICU and hospital stay, unplanned admission to ICU, and quality of recovery (QoR-15). We will use the following definitions:

- 1. Death: all-cause mortality at 90 days, then up to 12 months after surgery
- 2. A composite (pooled) and individual septic complications: sepsis, surgical site infection, anastomotic leak, and pneumonia
- 3. Sepsis: using Centers for Disease Control and Prevention (CDC) with National Healthcare Safety Network (NHSN) criteria:(72): two or more features of the systematic inflammatory response syndrome (SIRS) plus **evidence of a source or site of infection** (can be positive blood culture or purulence from any site):
  - i) Core temperature > 38°C or <36°C (core temperature was rectal or tympanic). If oral, inguinal or axillary temperatures were used, 0.5°C to be added to the measured value
  - ii) Heart rate > 90 beats per minute. If patient had an atrial arrhythmia, record the ventricular rate. If patients have a known medical condition or are receiving treatment that would prevent tachycardia (for example, heart block or beta blockers), they must meet two of the remaining three (a,b,c) SIRS criteria
    - a) Respiratory rate > 20 breaths per minute
    - b)  $PaCO_2 < 32 \text{ mmHg } (4.3 \text{ kPa})$
    - c) mechanical ventilation for an acute process
  - iii) White cell count of >12,000 mm<sup>3</sup> or < 4,000 mm<sup>3</sup>
- 4. Surgical site infection: using CDC criteria (http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf):
  - i) Superficial This includes one or more of the following:

- (1) purulent drainage from the superficial incision,
- (2) organisms isolated
- (3) diagnosis by surgeon or other physician or one of the signs or symptoms of infection- (pain or tenderness, localised swelling, redness or heat, superficial incision and is deliberately opened by surgeon.) (Unless culture negative)
- ii) Deep Incisional This includes one of the following:
  - (1) Purulent discharge from deep incision but not from organ/space component of the surgical site
  - (2) A deep incision spontaneously dehisces or is deliberately opened by surgeon with one addition sign (Temperature >38°C, localised pain, tenderness)
  - (3) An abscess or other evidence of infection
  - (4) Diagnosis by surgeon or other physician
- iii) **Organ/space** Occurred within 30 days with no implant or within 1 year if an implant is in place this includes one or more of the following
  - (1) Purulent discharge
  - (2) Organisms identified
  - (3) Abscess or evidence of infection involving the organ/space on examination
  - (4) Diagnosis by surgeon or other physician
- 5. **Pneumonia:** The presence of new and/or progressive pulmonary infiltrates on chest radiograph plus <u>two</u> or more of the following:
  - (1) Fever ≥ 38.5°C or postoperative hypothermia <36°C
  - (2) Leukocytosis ≥ 12,000 WBC/mm<sup>3</sup> or leukopenia < 4,000 WBC/mm<sup>3</sup>
  - (3) Purulent sputum and/or
  - (4) New onset or worsening cough or dyspnoea.
- 6. **Anastomotic leak:** A defect of the intestinal wall at the anastomotic site (including suture and staple lines of neorectal reservoirs) leading to a communication between the intra- an extra luminal compartments.
  - (1) Grade A anastomotic leakage results in no change in patients' management
  - (2) Grade B leakage requires active therapeutic intervention but is manageable without re- laparotomy
  - (3) Grade C anastomotic leakage requires re-laparotomy
- 7. Acute kidney injury: according to The Kidney Disease: Improving Global Outcomes (KDIGO) group criteria, but not urine output for Stage 2 or worse AKI defined as at least 2-fold increase in creatinine, or estimated GFR decrease >50%.(73) We also plan to report renal replacement therapy up to 90 days after surgery. Because a restrictive IV fluid regimen may artificially elevate serum creatinine due to a smaller dilutional effect from less IV fluids, we therefore calculated adjusted creatinine by first estimating the volume of distribution for creatinine as equal to total body water (assumed to be 60% of body weight, expressed in mL), and assuming that 50% of IV fluid was still accumulated as tissue oedema at the time of postoperative creatinine measurements.(74, 75) That is:

adjusted  $Cr = SCr \times (1 + [0.5 \times fluid\ balance/total\ body\ water])$ 

- 8. Pulmonary oedema: respiratory distress or impaired oxygenation AND radiological evidence of pulmonary oedema
- 9. Duration of mechanical ventilation: additive, for all episodes up to 90 days after surgery
- 10. Inflammation: plasma C-reactive protein (CRP, using site-specific assay) concentration on Day 3
- 11. Tissue perfusion: peak serum lactate within 24 hours of surgery
- 12. **Any blood transfusion:** including red cell, fresh frozen plasma or platelet transfusion, from the commencement of surgery
- 13. Unplanned admission to ICU within 30 days of surgery
- 14. Total ICU stay: additive, including initial ICU admission and readmission times up to Day 30
- 15. **Hospital stay:** additive, from the start (date, time) of surgery until actual hospital discharge , plus readmission(s) up to Day 30
- 16. Quality of recovery: QoR-15 score(76) on days 1, 3, and 30.
- 17.

Excessive fluid resuscitation can cause haemodilution (64) and dilutional coagulopathy, and this may increase the need for red cell and other blood transfusion (32). Blood transfusion is, of itself, associated with increased rates of sepsis and other postoperative complications (3, 24). All patients will have the same red cell transfusion trigger of 70 g/L, but this can be modified after assessment of cardiovascular risk (77, 78) or concern for active bleeding. Normal Saline, containing 154 mmol of sodium and 154 mmol of chloride per litre, is non-physiological and can lead to hyperchloraemic acidosis (33) and perhaps poorer outcome (79, 80). We will use a balanced salt solution as the routine fluid therapy in this study. The questionable value of urine output as a measure of kidney or other tissue perfusion will be emphasized (81).

Our study Group fluid regimens are aimed at distinct volume differences and according to recent recommendations (4, 72). The group-assigned fluid regimens will continue for at least 24 hours after surgery, or until cessation of IV fluid therapy (whichever occurs first). If the patient's clinical condition warrants modification to the type or rate of fluid administration, then such modifications can be made immediately. This does NOT imply that the patient is removed from the trial because we will analyze according to the intention-to-treat principle, but we will collect such data for secondary per-protocol and sensitivity analyses.

#### **Management of Oliguria**

It is a normal response of the body to attempt to conserve fluid in times of physiological stress. Oliguria (low urine output) is part of this homeostatic mechanism; there is no evidence it is harmful in the short term (first 24-48 h after surgery is common and not abnormal) (81). Nor is there any evidence that diuretics protect against AKI (82). We will however provide guidance to ward medical and nursing staff (see Procedures Manual).

#### 4. Experimental control

# 4.1 Group assignment

This will be a large, randomized, parallel-group, controlled trial. After stratification by centre and planned ICU/HDU admission (or not), patients will be randomly assigned from a computer-generated list (1:1) to either a Restrictive or Liberal fluid Group.

A 24-hr interactive voice recognition system (IVRS) will be available. An alternative web-based randomisation service will also be available during the conduct of the trial.

This is an intention to treat trial. Any participant who is randomised will be followed for the duration of the trial (unless they withdraw consent) even if they are withdrawn from the active phase of the trial. Patients who do not complete the active phase of the study will not be replaced.

## **Liberal Protocol**

The Liberal protocol group reflects common contemporary practices in Australia(29, 82), and is consistent with previous international trials (20, 24, 83) – see Appendix. At the commencement of surgery a bolus of Hartmann's balanced salt crystalloid 10 ml/kg followed by 8 ml/kg/h will be administered until the end of surgery – the latter can be further down-titrated after 4 hours if clinically indicated. Important: for the purposes of calculations of bolus and maintenance fluids in patients exceeding 100 kg, the maximal body weight will be set at 100 kg. A maintenance infusion will then continue at 1.5 ml/kg/h, for at least 24 hours, but this can be reduced postoperatively if there is evidence of fluid overload and no hypotension, and increased if there is evidence of hypovolaemia or hypotension. Alternative fluid types (crystalloid, dextrose, colloid) and electrolyte supplements will be allowed postoperatively in order to account for local preferences and patient biochemistry, for which we will collect data. For a 75-kg adult, the intraoperative volume (for a 4 h operation) will be 3150 ml (+colloid/blood replacement for blood loss), and then around 2700 ml per day. That is, the first (intraoperative + postoperative) 24-h fluid administration will be about 5400 ml (P.T.O).

## **Restrictive Protocol**

The Restrictive protocol group is designed to provide less than 2.0 L water and 120 mmol sodium per day. Induction of anaesthesia will be accompanied by an IV fluid bolus limited to ≤5 ml/kg; no other IV fluids will be used at the commencement of surgery (unless indicated by goal-directed device [see below]). Hartmann's balanced salt crystalloid 5 ml/kg/h will be administered until the end of surgery, and bolus colloid/blood used intraoperatively to replace blood loss (ml for ml); then an infusion at 0.8 ml/kg/h until expedited cessation of IV fluid therapy within 24 hours. The rate of postoperative fluid replacement can be reduced if there is evidence of fluid overload and no hypotension, and can

be increased if there is hypotension AND evidence of hypovolaemia. For a 75-kg patient and 4 h operation, intraoperative fluid volume will be 1875 ml (+colloid/blood replacement for blood loss). The first 24-h fluid administration will be around half that of the liberal group (P.T.O).



Hypotension will be initially treated with fluid boluses in the liberal protocol group, and with a vasoconstrictor in the restrictive protocol group. The latter will consist of metaraminol or phenylephrine bolus/infusion and/or noradrenaline infusion during surgery, and a noradrenaline infusion postoperatively if in a HDU or ICU environment. The lower limit of acceptable sBP in the restrictive group can be further reduced by the attending anaesthetist or intensivist in order to limit fluid replacement or potentially unnecessary inotropic support (as per above). We have laminated instructional flowcharts for the anaesthetists and postoperative (ward or ICU/HDU) medical and nursing staff caring for the study patients (see Appendix). Research staff will be present at or soon after all handover steps, and be contactable at all hours.

# 4.2 Goal-directed Therapy

For anaesthetists employing advanced monitoring (eg. CVP or goal-directed device), we allow additional colloid fluid supplementation to augment a haemodynamic target. It is likely to lead to additional colloid administration during and after surgery (3, 4, 45). Some hospitals use pulse contour analysis to direct perioperative or ICU fluid therapy in surgical patients, and some use oesophageal Doppler. Most rely upon conventional monitoring (HR, BP, urine output). We plan to test the effectiveness of each approach according to their local availability and use. The statistical analysis will focus

on a test for interaction, to determine whether the effects of a fluid regimen work differently in those with and without any advanced monitoring. We anticipate that more than half will use (only) clinical measures.

For each of the goal-directed techniques, pulse/stroke volume variation or FTc will be measured before commencement of surgery and repeated at regular (say, 10-30 min) intervals intraoperatively. For those in the liberal protocol group, goal-directed therapy can continue postoperatively at 4 hourly intervals, for up to 24 hours after surgery. If there is evidence of fluid responsiveness (eg. systolic pressure/volume variation of ≥13% (77)) at any of these times then IV colloid or crystalloid 3-5 ml/kg can be given. Such data will be collected on the CRF.

| Colloid* (recommended) or crystalloid (3 ml/kg) | Liberal | Restrictive |
|---|---|---|
| Colloid/blood (using a transfusion threshold) bolus if acute bleeding | Yes | Yes |
| If normotensive but monitoring suggests hypovolaemia (eg. CVP<5 or oliguria) | Yes | No |
| If normotensive but goal-directed device suggests hypovolaemia (eg. FTc <0.33, ΔSV ≥10%, or SVV≥13%) | Yes | Consider |
| If hypotensive (1) and hypovolaemia | Colloid* | Colloid* (but limit) + vasoconstrictor |
| (2) but not hypovolaemic | Colloid* ± vasoactive | vasoactive therapy |

<sup>\*</sup> starch-based colloids are not recommended (30, 34)

# 4.3 Blinding Procedure

Patients will be blinded to Group allocation. Anaesthetists, surgeons, and intensivists will have knowledge of Group identity. Similarly, it is expected that other surgical and nursing staff, and research staff conducting the in-hospital daily reviews, cannot be properly blinded to Group identity. But research staff conducting 1-12 mth follow-ups MUST be blinded to Group allocation.

#### **4.4 Case Report Forms**

For each form on which information is entered, the patient's initials, allocation number and the date of the visit must be entered in the appropriate space. The CRFs must be neatly handwritten with a black-ink ballpoint pen. Errors must be corrected by drawing a single line through the incorrect entry and writing in the new value positioned as close to the original as possible.

The correction must then be initialled and dated by the authorised individual making the change. Do not obliterate, write over, or erase the original entry when making a correction.

Case report forms should be opened as soon as possible following the start of screening and kept up to date as the patient continues the study.

As soon as possible after the end of each patient's participation in the study the CRF must be completed. All centres must store the paper based CRF according to GCP/ICP guidelines.

# 4.5 Web-based data entry

Following completion of the paper-based CRF, data will need to be entered by research staff to the database through a web-based data entry system. Further information can be found in the Procedures Manual. The system will audit the timeliness of data entry and reports will be generated the data monitoring committee regularly.

# 4.6 Data Base Production and Verification

Study data will be collected via the internet, monitored by the trial data management centre where all data fields are checked and automatically downloaded onto a database. At the end of the trial site-specific data will be sent to each site investigator on a CD, for long-term storage.

Study data will be collected in a paper based CRF, for transcription onto a web-database. We will maximize data quality and protocol standardization by arranging a start-up meeting at local scientific meetings or live streamed web based sessions, and will provide regular feedback to each centre via phone and the trial web-site, along with a monthly newsletter. A complete procedures manual will be produced. All study personnel will have 24-h access to the study coordinating centre to resolve any questions that arise. Further information can be found in the Procedures Manual.

# 4.7 Compliance Checks

Random audits of centres will be undertaken, to access the accuracy and legitimacy of the trial data. Statistical monitoring of the data completeness, data variance, and risk-appropriate endpoint rates will be done for all patient data.

## 4.8 Patient Completion/Withdrawal

All participants who are randomised will and undergo GA for surgery must be followed for the duration of the study (unless they withdraw consent) even if they are withdrawn from the active phase of the trial.

## 4.9 Repeat and Special Laboratory Tests

Serum electrolytes, haemoglobin/haematocrit, and a 12 lead ECG will be ordered preoperatively and if clinically indicated after surgery. All diabetics should have their HbA1C measured before surgery. Further tests will be ordered if clinically indicated.

#### **4.10 Adverse Experiences**

Serious adverse effects, serious adverse reactions, or suspected unexpected serious adverse reactions (SUSARs) are serious adverse events judged to be related to therapy.

At each visit/assessment, all adverse experiences either observed by the investigator or one of the clinical staff, or reported by the patient spontaneously <u>or</u> in response to a direct question will be evaluated by the investigator and noted in the adverse experience section of the patient's CRF. The nature of each experience, time of onset after surgery, duration, severity and relationship to treatment will be established. Any corrective treatment should be recorded on the appropriate pages of the CRF.

Adverse events should be documented at each assessment point throughout the study. Maximum intensity should be assigned to one of the following categories:

<u>Mild</u> - an adverse event which is easily tolerated by the patient, causing minimal discomfort and not interfering with everyday activities.

Moderate - an adverse event which is sufficiently discomforting to interfere with normal everyday activities.

<u>Severe</u> - an adverse event which is incapacitating and prevents normal everyday activities and/or requires therapeutic intervention (i.e. use of a prescription drug or hospitalisation).

Any serious adverse event should be reported by the local site investigator or research assistant within 24 hours by telephone or email to the local site investigator. Note that study endpoints <u>do not</u> need to be included as serious adverse events.

A preliminary telephone report should be followed by a full report which includes copies of relevant hospital case records, autopsy reports and other documents, where applicable.

A serious adverse experience is defined as any event which is fatal, life-threatening, permanently disabling or incapacitating or results in hospitalisation, prolongs a hospital stay or is associated with congenital abnormality, carcinoma or overdose.

<u>Life threatening</u> means that the patient was at immediate risk of death from the event as it occurred, ie. it does not include a reaction that, had it occurred in a more serous form, might have caused death. For example, drug induced hepatitis that resolved without evidence of hepatic failure would not be considered life threatening, even though drug induced hepatitis can be fatal.

<u>Permanent disability</u> means a permanent and substantial disruption of a patient's ability to carry out normal life functions.

More details for Adverse Event reporting will be found in the procedures manual.

#### 5. BIAS CONTROL

This is a large trial, randomised with permuted blocks (by centre and ICU). Anaesthetists, surgeons, and intensivists will have knowledge of Group identity. Similarly, it is expected that other surgical and nursing staff, and research staff conducting the in-hospital daily reviews, cannot be properly blinded to Group identity. But research staff conducting Day 3, 1-12 mth follow-ups MUST be blinded to Group allocation. Secondary outcomes are clearly defined in the protocol; disputes will be resolved by blinded assessors (endpoint adjudication committee).

#### 6. SAMPLE SIZE AND STATISTICAL ANALYSIS

All statistical analysis will be overseen by Prof Andrew Forbes, Monash University Department of Epidemiology and Preventive Medicine. The intention-to-treat population will include all patients randomly assigned to groups AND undergoing induction of anaesthesia.

Our initial sample size calculation was based primarily on our own data and other published studies. Our ENIGMA-II trial (n>5000 enrolled to date), with a lower risk study population, has a disability-free survival rate of 70% (15% mortality, 15% new disability) at 1 year after surgery). The most recent large data comes from the UK, where the 1-year mortality for open colorectal surgery was 17% in the 31,847 patients with pre-existing comorbidity (84). Reductions in serious complication rates have exceeded 25% in pooled analyses of similar studies(3, 82), and pre-existing major comorbidity increases mortality risk up to 16-fold (83). Using a type I error of 0.05 and survival analysis, with an expected one year disability-free survival probability of 65% (65) and a hazard ratio of ≥1.25, 1300 patients in each group will provide 90% power. Target recruitment was set at 2800 patients to account for losses due to follow-up. The Trial Steering Committee met on the 30<sup>th</sup> June, 2016, to discuss the results of a data quality committee review and statistician's report of the accruing incidence of disability. With near-complete information on 2,578 enrolled patients there were 300 events (disability or death); that is, a 12-month event rate of 14.6% - this is lower than expected. An increase in the trial sample size to 3,000 (≈380 events), which provides 80% power to detect HR≤0.75. This protocol amendment was accepted by the Steering Committee.

Analyses will be intention-to-treat. For analysis of the composite death-disability endpoint, we will use the Cox proportional hazards regression model with treatment as the only covariate to produce an unadjusted hazard ratio with a 95% confidence interval, together with Kaplan-Meier survival curves for graphical display; Analysis of secondary outcomes measured on a binary scale will be performed using log-binomial regression to estimate risk ratios with 95% confidence intervals, or exact logistic regression to approximate risk ratios if the number of events in either arm is fewer than 10. Time to event outcomes will use Cox proportional hazards regression as above. For analysis of the primary composite death-disability endpoint we will use the Cox proportional hazards regression model with treatment as the only covariate to produce an unadjusted hazard ratio with a 95% confidence interval, together with Kaplan-Meier survival curves for graphical display.

Outcomes measured on a continuous scale with a right skewed distribution will be log transformed and analysed using linear regression with robust standard errors, and outcomes with a left skewed distribution will be analysed with median regression with standard errors estimated using 1000 bootstrap replications.

# **Sensitivity Analysis**

Sensitivity analyses for all outcomes will use regression models with additional adjustment for the stratification variables of site and planned HDU/ICU destination status, plus any variables exhibiting substantial imbalance across treatment arms at baseline.

Sensitivity to missing outcome data will be performed using multiple imputation if the proportion of missing outcome data is greater than 5%. This will use baseline and auxiliary post-baseline information to inform the imputations under a *missing at random* assumption.

Planned sub-group analyses will assess patient sex, age groups (approximate quintiles), country, bowel surgery (yes/no), and use of any goal-directed techniques (yes/no). The latter include invasive or non-invasive cardiac output, stroke volume or pulse pressure variation, and oesophageal Doppler; but <u>not</u> include CVP monitoring. For these we will undertake tests for interaction by adding treatment-by-covariate terms to the regression models.

Additional prespecified subgroups will be tested for heterogeneity of effect, and their results considered exploratory (only): country, body mass index (BMI) categories (underweight, normal, overweight, obese, ≥super obese), ASA physical status (1/2, 3, 4), planned HDU/ICU destination status, and duration of surgery (approximate quintiles).

#### 7. INTERIM ANALYSIS

Interim analyses will consider the defined study endpoints, but include a specific consideration of 90-day mortality (because the primary endpoint is not finalised until 1 year after study entry) after enrolment of 1,445 patients, using the boundaries of O'Brien and Fleming. Results will be made available to the Data and Safety Monitoring Committee.

#### 8. SECONDARY ANALYSIS

We plan several substudies (to be funded from other sources), each of which will have a separate protocol and authorship plan (using an expanded list of contributors). Additional blood tests and other investigations will be done at selected hospitals according to local interest and expertise.

- 8.1 Cost-effectiveness, to include hospital stay and complications as we have done previously (85)
- **8.2** Hyperchloraemic acidosis (to measure strong ion difference, Cl-, lactate, albumin)
- **8.3** Pulmonary oedema (to measure FiO2/PaO2 ratio, CT/CXR-confirmed atelectasis)
- 8.4 Coagulopathy (to measure blood loss, platelet count, fibrinogen, INR, APTT, Hb flux, transfusion)
- **8.5** Sepsis (to measure fever, WCC, CRP and possibly other biomarkers)
- 8.6 AKI and hepatic injury
- 8.7 Postoperative cognitive deficit
- 8.8 Feeding and return of bowel function
- 8.9 Wound healing and anastomotic leak

# 9. PERSONNEL RESPONSIBILITIES

# 9.1 Investigators

The Steering Committee will consist of the principal investigator (PSM [Chair]), and other clinician-researchers in anaesthesia, surgery and intensive care medicine, plus the trial statistician – see below.

Each site investigator must ensure that all staff conducting the study are qualified to do so.

Each site investigator must submit the study protocol to the Ethics Committee or equivalent regulatory body and obtain approval prior to commencing the study.

Each site investigator must ensure that all staff involved with the study are fully instructed on the study procedures and are given access to the study protocol and other information relating to the study.

Each site investigator must ensure that the study is conducted in accordance with this protocol, ICH GCP notes for Guidance on Good Clinical Practice (CPMP/ICH/135/95) and in Australia with the NHMRC National Statement on Ethical Conduct in Research Involving Humans.

It is each site investigator's responsibility to ensure that written, informed consent is obtained from each patient prior to entering the study.

Each site investigator must ensure that the web-based CRFs are complete and accurate on completion of the study. Each site investigator will ensure that the quality control procedures are performed on both the CRFs and the data base.

It is the principal investigator's responsibility, in conjunction with the chief investigators, to write the Study Report at the completion of the study. Authorship guidelines are described in Section 11.

# 9.2 Monitor

Not applicable.

## 9.3 Sponsor

Alfred Health, as an investigator initiated study.

# 9.4 Steering Committee

The steering committee will include Paul Myles (chair), Rinaldo Bellomo, Tomas Corcoran, Chris Christophi, Andrew Forbes, Phil Peyton, David Story,, Kate Leslie, Jonathan Serpell, Shay McGuinness, Rachel Parke and Sophie Wallace (trial manager)

## 9.5 Endpoint Adjudication Committee (EAC)

Confirmation reports of all detected outcomes will be de-identified and re-labelled with study number. The committee will consist of experienced perioperative physicians. Details are provided in the Procedures Manual. Their role will be to resolve any uncertainty as to any of the above outcomes: additional advice can be sought by consultation with subspecialists.

#### 10. DATA SAFETY MONITORING COMMITTEE

The committee consists of Prof Monty Mythen (Chair, *intensivist*, Smiths Medical Professor of Anaesthesia & Critical Care, University College London (UK); Co-Director, Surgical Outcomes Research Centre), Prof Russell Gruen (*surgeon*, Professor of Surgery and Public Health, The Alfred & Monash University Director, National Trauma Research Institute; Melbourne), Prof John McNeil (*epidemiologist and triallist*, Professor of Epidemiology and Preventive Medicine; Head, School of Applied Clinical and Public Health Sciences; Monash University), Prof Guy Ludbrook (*anaesthetist*, Professor of Anaesthesia, Flinders University), and Dr Katherine Lee (*independent statistician*, MCRI).

The DMSC will discuss the interim results and vote for continuation or stopping the trial. A majority vote to stop the trial will be communicated to the Steering Committee at the Trial Coordinating Centre according to predetermined stopping rules (as above) and consideration of other relevant evidence. Their conduct is to be guided by the paper by DeMets et al. (86). Further details are provided in the DSMC charter.



# 11. ADMINISTRATIVE PROCEDURES

#### 11.1 Amendments to the Protocol

All modifications of the study will be written and filed as amendments to this protocol, maintaining original section identification. Such modification(s) will be made by the principal investigator, with endorsement by the Steering Committee and with the approval of the Ethics Committee (where applicable).

Any modifications to the study will be applied for all subsequent patients

#### 11.2 Early Termination or Extension of the Study

The investigator (with Ethics Committee approval) may discontinue or extend the study at any time.

## 11.3 Confidentiality/Publication of Study Results

Interim and preliminary results should not be discussed or presented outside the Trial Group, unless authorised by the chair of the Trial Steering Committee. The investigators plan to publish the results in a peer-reviewed journal.

#### 11.4 Retention of Records

All CRFs and all other documents associated with this study must be archived for at least 7 years following the completion of the trial, in accordance with TGA requirements.

#### 11.5 Audits

For the purpose of compliance with ICH GCP notes for Guidance on Good Clinical Practice (CPMP/ICH/135/95), it may be necessary for a regulatory agency to conduct a site audit.

Random audits may be conducted throughout the trial at the discretion of the Trial Steering Committee.

#### 12. ETHICAL PROCEDURES

#### 12.1 Guidelines for Good Clinical Practice

This study is to be performed in accordance with ICH GCP notes for Guidance on Good Clinical Practice (CPMP/ICH/135/95).

#### 12.2 Precautionary Advice

None specifically required.

# 12.3 Participant Information Sheet and Consent Form

The investigator or delegate will explain the study verbally to the patient. The patient will then be given a copy of the PI&CF and given an opportunity to read it and ask any questions of the investigator. The patient will be encouraged to obtain additional information about the study from an independent source. Once the patient is satisfied with the information they have received, has had an opportunity to ask questions and obtain additional information, and the investigator is satisfied that the patient truly understands the nature of the study, the patient will be asked to sign the consent form.

The signing of the consent form must take place in front of a witness and that witness must also be satisfied that the patient has a good understanding of the study. Each patient's signed consent form will be retained by the investigator.

Patients will be advised that they are free to refuse to participate in, or to withdraw from the study at any time. The medical care provided will not be affected by agreement or refusal to participate in this study. The original Consent Form for each subject will be stored in the Investigators file and a copy of the consent form will be placed in the patient's medical record.

# 12.4 Ethics Committee

This protocol will be submitted to the Ethics Committee (or relevant regulatory body) at each site and their approval obtained.

#### 13. AUTHORSHIP PLAN

# RELIEF Trial Authorship & Agreement

Target Journal: Lancet, New England Journal of Medicine, or JAMA

**Planned Authorship:** The RELIEF Trial Investigators

The trial will be described as a collaboration of the Australian and New Zealand College of Anaesthetists (ANZCA) Trials Group and the Australian and New Zealand Intensive Care Society (ANZICS) Clinical Trials Group.

The planned writing committee will include Paul Myles, Rinaldo Bellomo, Tomas Corcoran, Andrew Forbes, Philip Peyton, David Story, Chris Christophi, Andrew Davies, Kate Leslie, and Jonathan Serpell. This list may be extended or altered, according to a majority vote of the Trial Steering Committee.

Committee members and Site investigators at centres recruiting more than 250 patients will be offered co-authorship on at least one of the secondary publications. A more extensive participation and higher rate of patient enrolment may support a claim for authorship on the main publication (above), subject to a majority vote of the Trial Steering Committee.

Following acceptance for publication, all co-investigators (site investigators at each centre) can have access to all trial data if they would like to plan secondary analysis (and follow-up publication or presentation). A separate protocol should be developed and will require approval by the Trial Steering Committee before the presentation is made or submitted for publication.

An **Authorship Agreement** document will be produced before commencement of the trial, and all site investigators will be asked to sign their acknowledgement of this.

All site investigators listed in the appendix of the final publication(s) can be considered an author and so can list the publication(s) on their CVs.

# **Agreement to Participation**

I have read the trial protocol and agree to conduct the study according to the procedures outlined, and in accordance with Good Clinical Research Practice (GCRP) guidelines. Any information related to this trial will be kept confidential until publication or presentation at a scientific meeting. I have read and accept the proposed authorship plan.

| Site Coordinator (print): | |
|---------------------------|---------|
| Signature: | Date:// |

## References

- 1. Myles P, Leslie K. Anaesthesia for major abdominal and urological surgery. Evidence-based Anaesthesia and Intensive Care [textbook] In: Møller A, Pederson T (eds). 2006:223-46.
- 2. SIGN. Postoperative management in adults. A practical guide to postoperative care for clinical staff. Scottish Intercollegiate Guidelines Network (SIGN). 2004;77.
- 3. Rahbari NN, Zimmermann JB, Schmidt T, Koch M, Weigand MA, Weitz J. Meta-analysis of standard, restrictive and supplemental fluid administration in colorectal surgery. Br J Surg. 2009;96(4):331-41.
- 4. Bundgaard-Nielsen M, Secher NH, Kehlet H. 'Liberal' vs. 'restrictive' perioperative fluid therapy--a critical assessment of the evidence. Acta anaesthesiologica Scandinavica. 2009;53(7):843-51.
- 5. Chong PC, Greco EF, Stothart D, Maziak DE, Sundaresan S, Shamji FM, et al. Substantial variation of both opinions and practice regarding perioperative fluid resuscitation. Canadian journal of surgery Journal canadien de chirurgie. 2009;52(3):207-14.
- 6. Hannemann P, Lassen K, Hausel J, Nimmo S, Ljungqvist O, Nygren J, et al. Patterns in current anaesthesiological peri-operative practice for colonic resections: a survey in five northern-European countries. Acta anaesthesiologica Scandinavica. 2006;50(9):1152-60.
- 7. Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, et al. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet (London, England). 2008;372(9633):139-44.
- 8. Australian Institute of Health and Welfare A. Australian hospital statistics 2007-08. 2009.
- 9. Shires T, Williams J, Brown F. Acute change in extracellular fluids associated with major surgical procedures. Annals of surgery. 1961;154:803-10.
- 10. Arkilic CF, Taguchi A, Sharma N, Ratnaraj J, Sessler DI, Read TE, et al. Supplemental perioperative fluid administration increases tissue oxygen pressure. Surgery. 2003;133(1):49-55.
- 11. Mythen MG, Webb AR. The role of gut mucosal hypoperfusion in the pathogenesis of post-operative organ dysfunction. Intensive care medicine. 1994;20(3):203-9.
- 12. Davies SJ, Wilson RJ. Preoperative optimization of the high-risk surgical patient. British journal of anaesthesia. 2004;93(1):121-8.
- 13. Holte K, Klarskov B, Christensen DS, Lund C, Nielsen KG, Bie P, et al. Liberal versus restrictive fluid administration to improve recovery after laparoscopic cholecystectomy: a randomized, double-blind study. Annals of surgery. 2004;240(5):892-9.
- 14. Boyd O, Grounds RM, Bennett ED. A randomized clinical trial of the effect of deliberate perioperative increase of oxygen delivery on mortality in high-risk surgical patients. Jama. 1993;270(22):2699-707.
- 15. Wilson J, Woods I, Fawcett J, Whall R, Dibb W, Morris C, et al. Reducing the risk of major elective surgery: randomised controlled trial of preoperative optimisation of oxygen delivery. BMJ (Clinical research ed). 1999;318(7191):1099-103.
- 16. Arieff Al. Fatal postoperative pulmonary edema: pathogenesis and literature review. Chest. 1999;115(5):1371-7.
- 17. Ruttmann TG, James MF, Aronson I. In vivo investigation into the effects of haemodilution with hydroxyethyl starch (200/0.5) and normal saline on coagulation. British journal of anaesthesia. 1998;80(5):612-6.
- 18. Ratner AJ, Lysenko ES, Paul MN, Weiser JN. Synergistic proinflammatory responses induced by polymicrobial colonization of epithelial surfaces. Proceedings of the National Academy of Sciences of the United States of America. 2005;102(9):3429-34.
- 19. Lassen K, Soop M, Nygren J, Cox PB, Hendry PO, Spies C, et al. Consensus review of optimal perioperative care in colorectal surgery: Enhanced Recovery After Surgery (ERAS) Group recommendations. Archives of surgery (Chicago, III: 1960). 2009;144(10):961-9.
- 20. Lobo DN, Bostock KA, Neal KR, Perkins AC, Rowlands BJ, Allison SP. Effect of salt and water balance on recovery of gastrointestinal function after elective colonic resection: a randomised controlled trial. Lancet (London, England). 2002;359(9320):1812-8.
- 21. Tambyraja AL, Sengupta F, MacGregor AB, Bartolo DC, Fearon KC. Patterns and clinical outcomes associated with routine intravenous sodium and fluid administration after colorectal resection. World journal of surgery. 2004;28(10):1046-51; discussion 51-2.
- 22. Corcoran TR, JEJ. Clarke, S. Myles, PS. Oh, KM. Perioperative fluid management strategies in major surgery: a stratified meta-analysis. under peer review. 2011.
- 23. Brandstrup B, Tonnesen H, Beier-Holgersen R, Hjortso E, Ording H, Lindorff-Larsen K, et al. Effects of intravenous fluid restriction on postoperative complications: comparison of two perioperative fluid regimens: a randomized assessor-blinded multicenter trial. Annals of surgery. 2003;238(5):641-8.
- 24. Nisanevich V, Felsenstein I, Almogy G, Weissman C, Einav S, Matot I. Effect of intraoperative fluid management on outcome after intraabdominal surgery. Anesthesiology. 2005;103(1):25-32.

- 25. Kabon B, Akca O, Taguchi A, Nagele A, Jebadurai R, Arkilic CF, et al. Supplemental intravenous crystalloid administration does not reduce the risk of surgical wound infection. Anesthesia and analgesia. 2005;101(5):1546-53.
- 26. MacKay G, Fearon K, McConnachie A, Serpell MG, Molloy RG, O'Dwyer PJ. Randomized clinical trial of the effect of postoperative intravenous fluid restriction on recovery after elective colorectal surgery. The British journal of surgery. 2006;93(12):1469-74.
- 27. Holte K, Foss NB, Andersen J, Valentiner L, Lund C, Bie P, et al. Liberal or restrictive fluid administration in fast-track colonic surgery: a randomized, double-blind study. British journal of anaesthesia. 2007;99(4):500-8.
- 28. Vermeulen H, Hofland J, Legemate DA, Ubbink DT. Intravenous fluid restriction after major abdominal surgery: a randomized blinded clinical trial. Trials. 2009;10:50.
- 29. Myburgh J, Cooper DJ, Finfer S, Bellomo R, Norton R, Bishop N, et al. Saline or albumin for fluid resuscitation in patients with traumatic brain injury. The New England journal of medicine. 2007;357(9):874-84.
- 30. Perner A, Haase N, Guttormsen AB, Tenhunen J, Klemenzson G, Aneman A, et al. Hydroxyethyl starch 130/0.42 versus Ringer's acetate in severe sepsis. The New England journal of medicine. 2012;367(2):124-34.
- 31. Myburgh JA, Finfer S, Bellomo R, Billot L, Cass A, Gattas D, et al. Hydroxyethyl starch or saline for fluid resuscitation in intensive care. The New England journal of medicine. 2012;367(20):1901-11.
- 32. Finfer S, Bellomo R, Boyce N, French J, Myburgh J, Norton R. A comparison of albumin and saline for fluid resuscitation in the intensive care unit. The New England journal of medicine. 2004;350(22):2247-56.
- 33. Scheingraber S, Rehm M, Sehmisch C, Finsterer U. Rapid saline infusion produces hyperchloremic acidosis in patients undergoing gynecologic surgery. Anesthesiology. 1999;90(5):1265-70.
- 34. Myburgh JA, Finfer S, Bellomo R, Billot L, Cass A, Gattas D, et al. Hydroxyethyl Starch or Saline for Fluid Resuscitation in Intensive Care. N Engl J Med. 2012.
- 35. Marik PE, Baram M, Vahid B. Does central venous pressure predict fluid responsiveness? A systematic review of the literature and the tale of seven mares. Chest. 2008;134(1):172-8.
- 36. Peyton PJ, Chong SW. Minimally invasive measurement of cardiac output during surgery and critical care: a meta-analysis of accuracy and precision. Anesthesiology. 2010;113(5):1220-35.
- 37. Noblett SE, Snowden CP, Shenton BK, Horgan AF. Randomized clinical trial assessing the effect of Doppler-optimized fluid management on outcome after elective colorectal resection. The British journal of surgery. 2006;93(9):1069-76.
- 38. Conway DH, Mayall R, Abdul-Latif MS, Gilligan S, Tackaberry C. Randomised controlled trial investigating the influence of intravenous fluid titration using oesophageal Doppler monitoring during bowel surgery. Anaesthesia. 2002;57(9):845-9.
- 39. Wakeling HG, McFall MR, Jenkins CS, Woods WG, Miles WF, Barclay GR, et al. Intraoperative oesophageal Doppler guided fluid management shortens postoperative hospital stay after major bowel surgery. British journal of anaesthesia. 2005;95(5):634-42.
- 40. Futier E, Constantin JM, Petit A, Chanques G, Kwiatkowski F, Flamein R, et al. Conservative vs restrictive individualized goal-directed fluid replacement strategy in major abdominal surgery: A prospective randomized trial. Archives of surgery (Chicago, III: 1960). 2010;145(12):1193-200.
- 41. Walsh SR, Tang T, Bass S, Gaunt ME. Doppler-guided intra-operative fluid management during major abdominal surgery: systematic review and meta-analysis. International journal of clinical practice. 2008;62(3):466-70.
- 42. Mowatt G, Houston G, Hernandez R, de Verteuil R, Fraser C, Cuthbertson B, et al. Systematic review of the clinical effectiveness and cost-effectiveness of oesophageal Doppler monitoring in critically ill and high-risk surgical patients. Health technology assessment (Winchester, England). 2009;13(7):iii-iv, ix-xii, 1-95.
- 43. Gopal S, Jayakumar D, Nelson PN. Meta-analysis on the effect of dopexamine on in-hospital mortality. Anaesthesia. 2009;64(6):589-94.
- 44. Pearse RM, Belsey JD, Cole JN, Bennett ED. Effect of dopexamine infusion on mortality following major surgery: individual patient data meta-regression analysis of published clinical trials. Critical care medicine. 2008;36(4):1323-9.
- 45. Davies SJ, Yates D, Wilson RJT. Dopexamine Has No Additional Benefit in High-Risk Patients Receiving Goal-Directed Fluid Therapy Undergoing Major Abdominal Surgery. Anesthesia & Analgesia. 2011;112(1):130-8.
- 46. Hamilton MA, Cecconi M, Rhodes A. A systematic review and meta-analysis on the use of preemptive hemodynamic intervention to improve postoperative outcomes in moderate and high-risk surgical patients. Anesthesia and analgesia. 2011;112(6):1392-402.
- 47. Challand C, Struthers R, Sneyd JR, Erasmus PD, Mellor N, Hosie KB, et al. Randomized controlled trial of intraoperative goal-directed fluid therapy in aerobically fit and unfit patients having major colorectal surgery. British journal of anaesthesia. 2012;108(1):53-62.
- 48. Bellamy MC. Wet, dry or something else? British journal of anaesthesia. 2006;97(6):755-7.
- 49. Varadhan KK, Neal KR, Dejong CH, Fearon KC, Ljungqvist O, Lobo DN. The enhanced recovery after surgery (ERAS) pathway for patients undergoing major elective open colorectal surgery: a meta-analysis of randomized controlled trials. Clinical nutrition (Edinburgh, Scotland). 2010;29(4):434-40.

- 50. Myles PS, Devereaux PJ. Pros and cons of composite endpoints in anesthesia trials. Anesthesiology. 2010;113(4):776-8.
- 51. Myles PS, Hunt JO, Fletcher H, Solly R, Woodward D, Kelly S. Relation between quality of recovery in hospital and quality of life at 3 months after cardiac surgery. Anesthesiology. 2001;95(4):862-7.
- 52. Myles PS, Weitkamp B, Jones K, Melick J, Hensen S. Validity and reliability of a postoperative quality of recovery score: the QoR-40. British journal of anaesthesia. 2000;84(1):11-5.
- 53. Leslie K, Troedel S, Irwin K, Pearce F, Ugoni A, Gillies R, et al. Quality of recovery from anesthesia in neurosurgical patients. Anesthesiology. 2003;99(5):1158-65.
- Herrera FJ, Wong J, Chung F. A systematic review of postoperative recovery outcomes measurements after ambulatory surgery. Anesthesia and analgesia. 2007;105(1):63-9.
- 55. Kluivers KB, Riphagen I, Vierhout ME, Brolmann HA, de Vet HC. Systematic review on recovery specific quality-of-life instruments. Surgery. 2008;143(2):206-15.
- 56. Amemiya T, Oda K, Ando M, Kawamura T, Kitagawa Y, Okawa Y, et al. Activities of daily living and quality of life of elderly patients after elective surgery for gastric and colorectal cancers. Annals of surgery. 2007;246(2):222-8.
- 57. Myles PS, Hunt JO, Nightingale CE, Fletcher H, Beh T, Tanil D, et al. Development and psychometric testing of a quality of recovery score after general anesthesia and surgery in adults. Anesthesia and analgesia. 1999;88(1):83-90.
- 58. Myles P, Smith J, Knight J, Cooper D, Silbert B, McNeil J, et al. Aspirin and Tranexamic Acid for Coronary Artery Surgery (ATACAS) Trial: Rationale and design. American Heart Journal. 2008;155(2):224-30.
- 59. Myles PS, Leslie K, Peyton P, Paech M, Forbes A, Chan MT, et al. Nitrous oxide and perioperative cardiac morbidity (ENIGMA-II) Trial: rationale and design. American heart journal. 2009;157(3):488-94.e1.
- 60. Myles PS, Bellomo R. A pivotal trial of fluid therapy for major abdominal surgery: need and equipoise. Critical care and resuscitation: journal of the Australasian Academy of Critical Care Medicine. 2011;13(4):278-80.
- 61. Prowle JR, Chua HR, Bagshaw SM, Bellomo R. Clinical review: Volume of fluid resuscitation and the incidence of acute kidney injury a systematic review. Critical care (London, England). 2012;16(4):230.
- Tunis SR, Stryer DB, Clancy CM. Practical clinical trials: increasing the value of clinical research for decision making in clinical and health policy. Jama. 2003;290(12):1624-32.
- 63. Myles PS. Why we need large randomized studies in anaesthesia. British journal of anaesthesia. 1999;83(6):833-4.
- Rigg JR, Jamrozik K, Myles PS, Silbert BS, Peyton PJ, Parsons RW, et al. Epidural anaesthesia and analgesia and outcome of major surgery: a randomised trial. Lancet (London, England). 2002;359(9314):1276-82.
- 65. Myles PS, Peyton P, Silbert B, Hunt J, Rigg JR, Sessler DI. Perioperative epidural analgesia for major abdominal surgery for cancer and recurrence-free survival: randomised trial. BMJ (Clinical research ed). 2011;342:d1491.
- 66. Hubner M, Schafer M, Demartines N, Muller S, Maurer K, Baulig W, et al. Impact of Restrictive Intravenous Fluid Replacement and Combined Epidural Analgesia on Perioperative Volume Balance and Renal Function Within a Fast Track Program. J Surg Res. 2010.
- 67. Bijker JB, van Klei WA, Kappen TH, van Wolfswinkel L, Moons KG, Kalkman CJ. Incidence of intraoperative hypotension as a function of the chosen definition: literature definitions applied to a retrospective cohort using automated data collection. Anesthesiology. 2007;107(2):213-20.
- 68. Warschkow R, Beutner U, Steffen T, Muller SA, Schmied BM, Guller U, et al. Safe and early discharge after colorectal surgery due to C-reactive protein: a diagnostic meta-analysis of 1832 patients. Annals of surgery. 2012;256(2):245-50.
- 69. Nunes BK, Lacerda RA, Jardim JM. [Systematic review and meta-analysis of the predictive value of C-reactive protein in postoperative infections]. Revista da Escola de Enfermagem da U S P. 2011;45(6):1488-94.
- 70. Ustun T, Kostanjesek, N, Chatterji, S, Rehm, J Measuring Health and Disability: Manual for WHO Disability Assessment Schedule (WHODAS 2.0). Geneva: World Health Organization; 2010.
- 71. Organisation WH. World Report on Disability. <a href="http://wwwwhoint/disabilities/world-report/2011/reportpdf">http://wwwwhoint/disabilities/world-report/2011/reportpdf</a>. 2011;Technical appendix C:287-94.
- 72. Horan TC, Andrus M, Dudeck MA. CDC/NHSN surveillance definition of health care-associated infection and criteria for specific types of infections in the acute care setting. American journal of infection control. 2008;36(5):309-32.
- 73. Khwaja A. KDIGO clinical practice guidelines for acute kidney injury. Nephron Clinical practice. 2012;120(4):c179-84.
- 74. Liu KD, Thompson BT, Ancukiewicz M, Steingrub JS, Douglas IS, Matthay MA, et al. Acute kidney injury in patients with acute lung injury: impact of fluid accumulation on classification of acute kidney injury and associated outcomes. Crit Care Med. 2011;39(12):2665-71.
- 75. Christelis N, Wallace S, Sage CE, Babitu U, Liew S, Dugal J, et al. An enhanced recovery after surgery program for hip and knee arthroplasty. Med J Aust. 2015;202(7):363-8.
- 76. Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013;118(6):1332-40.

- 77. Hebert PC, Wells G, Blajchman MA, Marshall J, Martin C, Pagliarello G, et al. A multicenter, randomized, controlled clinical trial of transfusion requirements in critical care. Transfusion Requirements in Critical Care Investigators, Canadian Critical Care Trials Group. The New England journal of medicine. 1999;340(6):409-17.
- 78. Hebert PC, Yetisir E, Martin C, Blajchman MA, Wells G, Marshall J, et al. Is a low transfusion threshold safe in critically ill patients with cardiovascular diseases? Critical care medicine. 2001;29(2):227-34.
- 79. Shaw AD, Bagshaw SM, Goldstein SL, Scherer LA, Duan M, Schermer CR, et al. Major complications, mortality, and resource utilization after open abdominal surgery: 0.9% saline compared to Plasma-Lyte. Ann Surg. 2012;255(5):821-9.
- 80. Yunos NM, Bellomo R, Hegarty C, Story D, Ho L, Bailey M. Association between a chloride-liberal vs chloride-restrictive intravenous fluid administration strategy and kidney injury in critically ill adults. Jama. 2012;308(15):1566-72.
- 81. Prowle JR, Liu YL, Licari E, Bagshaw SM, Egi M, Haase M, et al. Oliguria as predictive biomarker of acute kidney injury in critically ill patients. Critical care (London, England). 2011;15(4):R172.
- 82. Zacharias M, Conlon NP, Herbison GP, Sivalingam P, Walker RJ, Hovhannisyan K. Interventions for protecting renal function in the perioperative period. The Cochrane database of systematic reviews. 2008(4):Cd003590.
- 83. Monk T, Saini V, Weldon B, Sigl J. Anesthetic management and one-year mortality after noncardiac surgery. Anesth Analg. 2005;100:4-10.
- 84. Mamidanna R, Burns EM, Bottle A, Aylin P, Stonell C, Hanna GB, et al. Reduced Risk of Medical Morbidity and Mortality in Patients Selected for Laparoscopic Colorectal Resection in England: A Population-Based Study. Arch Surg. 2011.
- 85. Graham AM, Myles PS, Leslie K, Chan MT, Paech MJ, Peyton P, et al. A cost-benefit analysis of the ENIGMA trial. Anesthesiology. 2011;115(2):265-72.
- 86. DeMets DL PS JD. The agonising negative trend in monitoring of clinical trials. Lancet (London, England). 1999(354):1983.